CLINICAL TRIAL: NCT01563055
Title: A Phase I/II, Open-label Study of Ofatumumab Added to Chlorambucil in Previously Untreated Japanese Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115601
Record Dates: First submitted 2012-03-15; First posted 2012-03-26 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Leukaemia, Lymphocytic, Chronic
MeSH Terms: conditions — Leukemia, B-Cell | interventions — Chlorambucil; Tablets; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ofatumumab + chlorambucil (Experimental): ofatumumab dose: cycle 1 300mg day 1 and 1000mg day 8, subsequent cycles: 1000mg at day 1 every 28 days; chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 treatment cycles
  Interventions: Drug: chlorambucil, tablets; Drug: ofatumumab (GSK1841157) infusion

INTERVENTIONS:
Drug: chlorambucil, tablets — 2mg tablets, chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 cycles
Drug: ofatumumab (GSK1841157) infusion — iv infusion; dose: cycle 1 300mg day 1 and 1000mg day 8, subsequent cycles: 1000mg at day 1 every 28 days;

SUMMARY:
This is an open-label study to evaluate tolerability, safety, efficacy and pharmacokinetic profile of ofatumumab in combination with chlorambucil in Japanese patients with previously untreated Chronic Lymphocytic Leukemia (CLL).

DETAILED DESCRIPTION:
This is an open-label study to evaluate tolerability, safety, efficacy and pharmacokinetic profile of ofatumumab in combination with chlorambucil in Japanese patients with previously untreated Chronic Lymphocytic Leukemia (CLL). Ofatumumab will be infused intravenously at Day 1 (300 mg) and Day 8 (1000 mg) in the first 28-day cycle, followed by infusions of 1000 mg at the first day of each 28-day cycle. Chlorambucil will be given 10 mg/m2 at Day 1-7 in each 28-day cycle.

The primary objectives are to evaluate tolerability and overall response rate (ORR) of ofatumumab with chlorambucil for previously untreated (frontline) CLL.

Secondary objectives include to evaluate complete remission (CR) rate, progression free survival (PFS), overall survival (OS), time to response, duration of response, time to next therapy, incidence and severity of adverse events and serious adverse events, incidences of grade 3 and 4 infections and myelosuppression (anemia, neutropenia, thrombocytopenia), and pharmacokinetics of ofatumumab and chlorambucil.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL defined by : Circulating B lymphocytes ≥5,000 /μL AND Flow cytometry confirmation of immunophenotype with CD5, CD19, CD20, and CD23 prior to Visit 2.
* Considered inappropriate for fludarabine-based therapy
* Active disease and indication for treatment based on modified NCI-WG guidelines defined by presenting at least any one of the following conditions :

Evidence of progressive marrow failure as manifested by development or worsening of anemia and/or thrombocytopenia.

Massive (i.e. at least 6 cm below the left costal margin) or progressive or symptomatic splenomegaly.

Massive nodes (i.e. at least 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.

Progressive lymphocytosis with an increase of more than 50% over a two month period or an lymphocyte doubling time of less than 6 months.

A minimum of any one of the following disease-related symptoms must be present : a) Unintentional Weight loss ≥ 10% within the previous six months ; b) Fevers >38.0 degree C for ≥ 2 weeks without evidence of infection ; or c) Night sweats for more than 1 month without evidence of infection.

* Not been previously treated for CLL (prior autoimmune hemolytic anemia treatment permitted).
* ECOG Performance Status of 0-2.
* Life expectancy of at least 6 months, in the opinion of the investigator.
* Age ≥ 20 years.
* Signed written informed consent prior to performing any study-specific procedures.
* Patients possible to stay at the trial site for at least two days (the day of the first infusion and a subsequent day).

Exclusion Criteria:

* Prior immuno- or chemotherapy for CLL or small lymphocytic lymphoma (SLL) with any agent except corticosteroids used to treat autoimmune hemolytic anemia.
* Previous autologous or allogeneic stem cell transplantation.
* Active autoimmune hemolytic anemia (AIHA) requiring corticosteroid therapy > 100 mg/day equivalent to hydrocortisone, or chemotherapy.
* Known transformation of CLL (e.g. Richter).
* Known CNS involvement of CLL.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to screening (Visit 1), congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities.
* History of significant cerebrovascular disease or event with significant symptoms or sequelae*.
* Glucocorticoid use, unless given in doses ≤ 100 mg/day hydrocortisone (or equivalent dose of other glucocorticoid) for <7 days for exacerbations other than CLL (e.g. asthma).
* Known HIV positive.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb and/or HBsAb positive, an HBV DNA test will be performed and if positive the subject will be excluded.
* Screening laboratory values :

Creatinine > 2.0 times upper normal limit (unless normal creatinine clearance). Total bilirubin > 2.0 times upper normal limit (unless due to Gilbert's syndrome).

Alanine transaminase (ALT) > 3.0 times upper normal limit.

* Previous treatment or known or suspected hypersensitivity to ofatumumab that in the opinion of the investigator or medical monitor is a contraindication to their participation in the present study.
* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to Visit 1, whichever is longer, treatment with any anti-CD20 monoclonal antibody within 3 months of Visit 1, or participation in any other interventional clinical study. Note: Participation in any other interventional clinical study after disease progression during post PD-follow-up is permitted.
* Known or suspected inability to comply with study protocol.
* Lactating women, women with a positive pregnancy test at Visit 1 or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception from study start through one year following last treatment dose. Adequate contraception is defined as oral hormonal birth control, intrauterine device, male partner sterilization (if male partner is sole partner for that subject) and the double barrier method (condom or occlusive cap plus spermicidal agent).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of two parts. In part A of the study, the eligible participants (par.) were enrolled to assess the tolerability of ofatumumab with chlorambucil. After confirmation of the tolerability, Part B of the study was initiated. The total number of participants in Part A and Part B was 10.
Groups:
- Ofatumumab + Chlorambucil: Par. with previously untreated chronic lymphocytic leukemia (CLL) received intravenous (IV) infusions of ofatumumab on Day 1 (300 milligrams [mg]) and Day 8 (1000 mg) in the first cycle, followed by 1000 mg on the first day of each subsequent 28-day cycle in combination with oral chlorambucil 10 mg/meter squared (m^2) on Days 1-7 of each cycle for at least 3 cycles, until best overall response or up to 12 cycles. After the Treatment Phase (for par. in CR, PR or SD), survival and disease status were assessed 28 days after the first day of the last treatment cycle (Follow-up [FU] 1), 84 and 168 days after the day of FU1 (FU85 and FU169, respectively). For par. with disease progression (PD) during the Treatment Phase, post PD follow-up were done 28 days after the first day of the last treatment cycle (PDFU1) to assess safety. Survival status, date of next CLL therapy, and type of therapy were subsequently assessed 84 and 168 days after the day of PDFU1 (PDFU85 and PDFU169, respectively).
Period: Overall Study
Arm/Group | Ofatumumab + Chlorambucil
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (10.38)
Age, Customized [Number; unit: Participants]
  <65 years | 1
  >=65 years | 9
  >=75 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Toxicity Requiring Discontinuation From Study Treatment During Cycle 1
Description: Tolerability of ofatumumab in combination with chlorambucil was evaluated based on the number of participants who developed toxicity requiring discontinuation from study treatment during Cycle 1. The treatment was considered tolerable when 0 of 3 participants, or <=2 of 6 participants developed toxicity which required discontinuation of study treatment during Cycle 1. The toxicity requiring discontinuation was determined based on the pre-defined withdrawal criteria.
Time Frame: From start of treatment through Cycle 1 (Week 4)
Population: All Subjects Population: all participants who received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Number of Participants With Overall Response, as Assessed by the Independent Review Committee (IRC) With CT, IRC and Investigator
Description: Response evaluated as per International Workshop for Chronic Lymphocytic Leukemia (IWCLL) National Cancer Institute-sponsored Working Group (NCI-WG) Guidelines, 2008. Overall response rate (ORR) is defined as percentage of par. achieving complete remission (CR), nodular partial remission (nPR), CR-incomplete (CRi) or PR. CR (>=2 months after last treatment): lymphocytes (LC) <4000 per microliter (μL), no lymphadenopathy (Ly)>1.5 cm/hepatomegaly/splenomegaly/constitutional symptoms; neutrophils (N)>1500/µL, platelets (PL)>100,000/µL, hemoglobin (Hb)>11 grams/deciliter (g/dL), bone marrow (BM) sample must be normocellular for age,<30% LC, no lymphoid nodule (LN). PR:>=50% decrease in LC, Ly, size of liver and spleen; and at least one of these: N>1500/μL, PL>100,000/µL or 50% improvement over Baseline (BL), Hb>11 g/dL or 50% improvement over BL. nPR: persistent nodules BM. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity.
Time Frame: From start of treatment until disease progression or death (up to Week 62.3)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  IRC with CT Assessed, CR | 0
  IRC with CT Assessed, CRi | 0
  IRC with CT Assessed, nPR | 0
  IRC with CT Assessed, PR | 5
  IRC Assessed, CR | 1
  IRC Assessed, CRi | 0
  IRC Assessed, nPR | 1
  IRC Assessed, PR | 5
  Investigator Assessed, CR | 1
  Investigator Assessed, CRi | 0
  Investigator Assessed, nPR | 0
  Investigator Assessed, PR | 6

3. Secondary Outcome: Number of Participants With CR, as Assessed by the IRC, IRC With CT, and the Investigator
Description: Response was determined according to the IWCLL updated NCI-WG guidelines, 2008. According to the guidelines, CR (all the criteria at least 2 months after last treatment): peripheral blood lymphocytes below < 4,000/μL, no Ly > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; Neu >1500 /µL, PL >100,000/µL, Hb >11 g/dL, BM sample must be normocellular for age, <30% lymphocytes, no LN. PR: >=50% decrease in peripheral blood lymphocytes, Ly, size of liver and spleen; and blood count showing at least one of the following results: Neu>1500/μL, PL >100,000/µL or 50% improvement over BL, Hb >11 g/dL or 50% improvement over BL. No increase in LN and no new LN.
Time Frame: From start of treatment until disease progression or death (up to Week 62.3)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  IRC with CT Assessed, CR | 0
  IRC Assessed, CR | 1
  Investigator Assessed, CR | 1

4. Secondary Outcome: Progression-free Survival (PFS), as Assessed by the IRC and the Investigator
Description: Progression free survival is defined as the time from start of treatment until disease progression (PD) or death due to any cause. PD was determined by the IRC or investigator according to the definitions of response in the IWCLL updated NCI-WG guidelines, 2008. According to the guidelines, PD is characterized by at least one of the following: lymphadenopathy (appearance of any new lesion such as enlarged lymph nodes (>1.5 centimeter [cm]), spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site); an increase by 50% or more in the previously noted enlargement of the liver or spleen; an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 per microliter B-lymphocytes; transformation to a more aggressive histology; or occurrence of cytopenia attributable to chronic lymphocytic leukemia. PFS was censored at the last visit with adequate assessment for participants who were alive and had not progressed.
Time Frame: From start of treatment until disease progression or death (up to Week 62.3)
Population: All Subjects Population. Only participants who progressed or died were analyzed.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Weeks
  IRC Assessed, Response, n=1 | NA [6.1 to NA] — No PFS could be determined because only one progression or death was observed in the participants, and other 9 participants were censored for analysis Not enough events to estimate upper limit of confidence interval
  Investigator Assessed, Response, n=1 | NA [16.1 to NA] — No PFS could be determined because only one progression or death was observed in the participants, and other 9 participants were censored for analysis Not enough events to estimate upper limit of confidence interval

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as time from start of treatment until death due to any cause. For participants who did not die, time to death was censored at the time of the last date of contact.
Time Frame: From start of treatment until death (up to Week 62.3
Population: All Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Weeks | NA [NA to NA] — All participants were alive at the time of the last follow-up and thus were censored for the analysis

6. Secondary Outcome: Time to Response, as Assessed by the IRC
Description: Time to response is defined as the time from start of treatment until the first response (CR/CRi/nPR/PR). Response was determined according to the IWCLL updated NCI-WG guidelines, 2008. This analysis only included participants who had a response while in the study, there was no censoring.
Time Frame: From start of treatment until the first response (CR/CRi/nPR/PR) (up to Week 62.3)
Population: All Subjects Population. Only those participants classified as responders (CR, CRi, PR, nPR) were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 7
Weeks | 4.1 [4.1 to 6.1]

7. Secondary Outcome: Duration of Response, as Assessed by the IRC
Description: Duration of response is defined as the time from the first documented evidence of CR, CRi, nPR or PR until the first documented sign of PD or death in participants with CR, CRi, nPR or PR. For participants who did not progress or die, duration of response was censored on the date of last assessment.
Time Frame: From initial response (CR/CRi/nPR/PR) until disease progression or death (up to Week 62.3)
Population: All Subjects Population. Only those participants classified as responders (CR, CRi, PR, nPR) were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 7
Weeks | NA [NA to NA] — The duration of response could not be assessed because no progression was observed in any of the participants.

8. Secondary Outcome: Time to Next Chronic Lymphocytic Leukemia (CLL) Therapy
Description: Time to next CLL therapy is defined as the time from start of treatment until the first administration of the next CLL treatment other than chlorambucil administrations scheduled in this study. Time to next CLL therapy was restricted to the subgroup of the population who receive a next CLL therapy after experiencing disease progression.
Time Frame: From start of treatment until the first administration of the next CLL therapy (up to Week 62.3)
Population: All Subjects Population. Only those participants who received next CLL therapy were evaluated.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 1
Weeks | 11.4 [NA to NA] — No 95% CI were available because only one participant received the next CLL therapy.

9. Secondary Outcome: Number of Participants With no B-symptoms (Constitutional Symptoms) and With at Least One B-symptom (Constitutional Symptoms) at the Indicated Time Points
Description: The number of participants with no B-symptoms (no night sweat [without signs of infection], no unexplained, unintentional weight loss >= 10% within the previous 6 months, no recurrent, unexplained fever of greater than 38 degrees celcius for 2 weeks and no extreme fatigue) and the number of participants with at least one of the B-symptoms are summarized by assessment time. The presence of the B-symptoms was assessed at Baseline, Day 1 of each treatment cycle and follow-up (FU). Baseline was the last pre-dose assessment performed at Cycle (C) 1-Day (D) 1.
Time Frame: Baseline, C2-D29, C3-D57, C4-D85, C5-D113, C6-D141, C7-D169, C8-D197, C9 -D225, FU 1-PDFU 1 (28 days post Day 1 of Last Cycle), FU 85-PDFU 85 (84 days after FU-1), and FU 169-PDFU 169 (168 days after FU-1)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  Baseline, With no B-symptom, n=10 | 9
  Baseline, With at least one B-symptom, n=10 | 1
  Cycle 2-Day 29, With no B-symptom, n=8 | 8
  Cycle 2-Day 29, With at least one B-symptom, n=8 | 0
  Cycle 3-Day 57, With no B-symptom, n=8 | 8
  Cycle 3-Day 57, With at least one B-symptom, n=8 | 0
  Cycle 4-Day 85, With no B-symptom, n=7 | 7
  Cycle 4-Day 85, With at least one B-symptom, n=7 | 0
  Cycle 5-Day 113, With no B-symptom, n=7 | 7
  Cycle 5-Day 113, With at least one B-symptom, n=7 | 0
  Cycle 6-Day 141, With no B-symptom, n=7 | 7
  Cycle 6-Day 141, With at least one B-symptom, n=7 | 0
  Cycle 7-Day 169, With no B-symptom, n=2 | 2
  Cycle 7-Day 169, With at least one B-symptom, n=2 | 0
  Cycle 8-Day 197, With no B-symptom, n=2 | 2
  Cycle 8-Day 197, With at least one B-symptom, n=2 | 0
  Cycle 9-Day 225, With no B-symptom, n=2 | 2
  Cycle 9-Day 225, With at least one B-symptom, n=2 | 0
  FU 1-PDFU 1, With no B-symptom, n=9 | 9
  FU 1-PDFU 1, With at least one B-symptom, n=9 | 0
  FU 85-PDFU 85, With no B-symptom, n=9 | 9
  FU 85-PDFU 85, With at least one B-symptom, n=9 | 0
  FU 169-PDFU 169, With no B-symptom, n=8 | 8
  FU 169-PDFU 169, With at least one B-symptom, n=8 | 0

10. Secondary Outcome: Number of Participants With Improvement in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS is a scale to assess disease progression, extent to which disease affects the daily living abilities and determines appropriate treatment and prognosis. It is scored on a scale of 0 to 5 as, 0 (fully active), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), 2 (ambulatory and capable of all self cares but unable to carry out any work activities, up and about > 50% of waking hours), 3 (capable of only limited self cares, confined to bed or chair > 50% of waking hours), 4 (completely disabled, cannot carry on any self cares, totally confined to bed or chair), 5 (death). Improvement is defined as decrease from Baseline by at least one step on the ECOG performance status scale (yes/no). Baseline was the last pre-dose assessment performed on Cycle 1-Day 1(C1-D1). When C1-D1 was missing, the last assessment performed prior to pre-dose C1-D1 was used. It was performed on Day 1 of each cycle and follow-up (FU).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  Cycle 2-Day 29, Improved, n=8 | 0
  Cycle 2-Day 29, No change, n=8 | 8
  Cycle 2-Day 29, Deteriorated, n=8 | 0
  Cycle 3-Day 57, Improved, n=8 | 0
  Cycle 3-Day 57, No change, n=8 | 8
  Cycle 3-Day 57, Deteriorated, n=8 | 0
  Cycle 4-Day 85, Improved, n=7 | 0
  Cycle 4-Day 85, No change, n=7 | 7
  Cycle 4-Day 85, Deteriorated, n=7 | 0
  Cycle 5-Day 113, Improved, n=7 | 0
  Cycle 5-Day 113, No change, n=7 | 7
  Cycle 5-Day 113, Deteriorated, n=7 | 0
  Cycle 6-Day 141, Improved, n=7 | 0
  Cycle 6-Day 141, No change, n=7 | 6
  Cycle 6-Day 141, Deteriorated, n=7 | 1
  Cycle 7-Day 169, Improved, n=2 | 0
  Cycle 7-Day 169, No change, n=2 | 2
  Cycle 7-Day 169, Deteriorated, n=2 | 0
  Cycle 8-Day 197, Improved, n=2 | 0
  Cycle 8-Day 197, No change, n=2 | 2
  Cycle 8-Day 197, Deteriorated, n=2 | 0
  Cycle 9-Day 225, Improved, n=2 | 0
  Cycle 9-Day 225, No change, n=2 | 2
  Cycle 9-Day 225, Deteriorated, n=2 | 0
  FU 1-PDFU 1, Improved, n=9 | 0
  FU 1-PDFU 1, No change, n=9 | 9
  FU 1-PDFU 1, Deteriorated, n=9 | 0
  FU 85-PDFU 85, Improved, n=9 | 0
  FU 85-PDFU 85, No change, n=9 | 8
  FU 85-PDFU 85, Deteriorated, n=9 | 1
  FU 169-PDFU 169, Improved, n=8 | 0
  FU 169-PDFU 169, No change, n=8 | 8
  FU 169-PDFU 169, Deteriorated, n=8 | 0

11. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed.
Time Frame: From start of treatment until follow-up for survival (up to Week 62.3)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  Any AE | 10
  Any SAE | 2

12. Secondary Outcome: Number of Participants With AEs of Maximum Severity
Description: Adverse events were graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) grade, version 4.03 (1=mild; 2=moderate; 3=severe; 4=life-threatening/disabling; 5=death). AEs not in the list of CTCAE were graded at discretion of the investigator.
Time Frame: From start of treatment until follow-up for survival (up to Week 62.3)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  Any AE Grade 1 | 0
  Any AE Grade 2 | 4
  Any AE Grade 3 | 5
  Any AE Grade 4 | 1
  Any AE Grade 5 | 0

13. Secondary Outcome: Number of Participants With the Indicated Grade 3 or Grade 4 Adverse Events
Description: Adverse events were graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) grade, version 4.03 (1=mild; 2=moderate; 3=severe; 4=life-threatening/disabling; 5=death). AEs not in the list of CTCAE were graded at discretion of the investigator. Myelosuppression is defined as the decrease in the ability of the bone marrow to produce blood cells. Participants with Grade (G)3 or G4 adverse event of infection and myelosuppression (anemia, neutropenia, and thrombocytopenia) are presented. Also presented are number of participants with autoimmune hemolytic anemia (AIHA). AIHA is a disease where the body's immune system fails to recognize red blood cells as "self" and begins destroying these red blood cells.
Time Frame: From start of treatment until follow-up for survival (up to Week 62.3)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  Infections, G3 | 0
  Infections, G4 | 0
  Thrombocytopenia, G3 | 2
  Thrombocytopenia, G4 | 0
  Neutropenia, G3 | 2
  Neutropenia, G4 | 1
  Anemia, G3 | 0
  Anemia, G4 | 0
  Autoimmune Hematologic Complication | 0

14. Secondary Outcome: Number of Participants With the Indicated Results for Human Anti-human Antibody (HAHA) at the Indicated Time Points
Description: HAHA are indicators of immunogenicity induced by ofatumumab. Blood samples were taken from participants at Screening, Cycle 4-Day 85, FU 1-PDFU 1, and FU 169-PDFU 169. The presence of HAHA in human serum was determined using a validated electrochemiluminescent assay in a multi-tier assay format. The results are presented as participants with HAHA results as positive, negative or confirmation required.
Time Frame: Screening, Cycle 4-Day 85, FU 1-PDFU 1 (28 days post Day 1 of Last Cycle), and FU 169-PDFU 169 (168 days after FU-1)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Participants
  Screening, Positive, n=10 | 1
  Screening, Negative, n=10 | 9
  Screening, Confirmation required, n=10 | 0
  Cycle 4-Day 85, Positive, n=7 | 0
  Cycle 4-Day 85, Negative, n=7 | 7
  Cycle 4-Day 85, Confirmation required, n=7 | 0
  FU 1-PDFU 1, Positive, n=10 | 0
  FU 1-PDFU 1, Negative, n=10 | 10
  FU 1-PDFU 1, Confirmation required, n=10 | 0
  FU 169-PDFU 169, Positive, n=8 | 0
  FU 169-PDFU 169, Negative, n=8 | 8
  FU 169-PDFU 169, Confirmation required, n=8 | 0

15. Secondary Outcome: Mean Change From Baseline in the Immunoglobulins (Ig) Antibodies IgA, IgG, and IgM at the Indicated Time Points
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants. Baseline IgA, IgG, and IgM values are the last pre-dose assessment values performed on Cycle 1-Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Immunoglobulins were measured at Cycle 1-Day 1, FU 1-PDFU 1, and FU 169-PDFU 169 for participants in CR, PR, and stable disease (SD).
Time Frame: Baseline (Cycle 1-Day 1), FU 1-PDFU 1 (28 days post Day 1 of Last Cycle), and FU 169-PDFU 169 (168 days after FU-1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Grams per liter
  IgA, FU 1-PDFU 1, n=10 | 0.111 (0.2816)
  IgA, FU 169-PDFU 169, n=8 | 0.326 (0.4172)
  IgG, FU 1-PDFU 1, n=10 | -0.025 (1.4555)
  IgG, FU 169-PDFU 169, n=8 | 0.611 (1.0636)
  IgM, FU 1-PDFU 1, n=10 | -0.053 (0.1466)
  IgM, FU 169-PDFU 169, n=8 | -0.045 (0.1466)

16. Secondary Outcome: Number of Participants Who Were Positive or Negative for Minimal Residual Disease (MRD), as Assessed by IRC With CT
Description: MRD refers to small number of leukemic cells that remain in the participant's body during treatment or after treatment in participants who achieved a confirmed complete remission. MRD assessment in bone marrow aspiration sample was perfrmed by flow cytometry (cluster of differentiation [CD]5, CD19, CD20, CD23). The absence of MRD was defined as less than one CLL cell per 10,000 leukocytes. The number of participants who were positive and negative for MRD are presented.
Time Frame: FU 85-PDFU 85 (84 days after FU-1)
Population: All Subjects Population. Only those participants who were positive and negative for MRD were analyzed.
Measure: Number; unit: Participants
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 8
Participants
  Positive | 4
  Negative | 4

17. Secondary Outcome: Change From Baseline in CD5+CD19+ and CD5-CD19+ Cell Counts at the Indicated Time Points
Description: CD5+CD19+ cells were counted in peripheral blood by flow cytometry. Baseline CD5+CD19+ and CD5-CD19+ cell count value is the last pre-dose assessment values performed on Cycle 1-Day 1. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. B-cell monitoring (CD5+CD19+ and CD5-CD19+) was performed at Cycle 1 (Day 1, Day 15) and Cycle 2 (Day 29, Day 43), on Day 1 of Cycle 3, 4, 5, 6, 9 and 12 (Day 57, Day 85, Day 113, Day 141, Day 225, Day 309), 28 days after the first day of the last treatment cycle (FU 1-PDFU 1) for all participants depending on the number of cycles administered, and 84 and 168 days after the day of FU 1-PDFU 1 for participants in CR, PR, and SD.
Time Frame: Baseline, C1-D15, C2-D29, C2-D43, C3-D57, C4-D85, C5-D113, C6-D141, C7-D169, C8-D197, C9-D225, FU 1-PDFU 1 (28 days post Day 1 of Last Cycle), FU 85-PDFU 85 (84 days after FU-1), and FU 169-PDFU 169 (168 days after FU-1)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Cells per microliter
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Cells per microliter
  CD5+CD19+, Cycle 1-Day 15, n=8 | -71066.50 (114877.018)
  CD5+CD19+, Cycle 2-Day 29, n=8 | -50441.25 (56969.080)
  CD5+CD19+, Cycle 2-Day 43, n=8 | -36755.88 (36719.313)
  CD5+CD19+, Cycle 3-Day 57, n=8 | -31823.50 (37479.968)
  CD5+CD19+, Cycle 4-Day 85, n=7 | -35679.00 (39379.825)
  CD5+CD19+, Cycle 5-Day 113, n=7 | -35754.71 (39502.575)
  CD5+CD19+, Cycle 6-Day 141, n=7 | -35791.43 (39535.868)
  CD5+CD19+, Cycle 7-Day 169, n=2 | -61591.00 (19469.478)
  CD5+CD19+, Cycle 8-Day 197, n=2 | -61589.00 (19473.721)
  CD5+CD19+, Cycle 9-Day 225, n=2 | -61591.00 (19470.892)
  CD5+CD19+, FU 1-PDFU 1, n=10 | -59868.20 (96360.514)
  CD5+CD19+, FU 85-PDFU 85, n=9 | -31370.78 (36239.779)
  CD5+CD19+, FU 169- PDFU 169, n=8 | -31270.25 (38733.484)
  CD19+CD5-, Cycle 1-Day 15, n=8 | -6752.50 (14473.357)
  CD19+CD5-, Cycle 2-Day 29, n=8 | -6616.13 (14070.593)
  CD19+CD5-, Cycle 2-Day 43, n=8 | -6044.00 (12496.749)
  CD19+CD5-, Cycle 3-Day 57, n=8 | -2867.13 (4561.234)
  CD19+CD5-, Cycle 4-Day 85, n=7 | -1792.57 (3669.425)
  CD19+CD5-, Cycle 5-Day 113, n=7 | -1792.43 (3668.705)
  CD19+CD5-, Cycle 6-Day 141, n=7 | -1794.14 (3668.713)
  CD19+CD5-, Cycle 7-Day 169, n=2 | -362.50 (64.347)
  CD19+CD5-, Cycle 8-Day 197, n=2 | -362.00 (63.640)
  CD19+CD5-, Cycle 9-Day 225, n=2 | -362.00 (63.640)
  CD19+CD5-, FU 1-PDFU 1, n=10 | -7534.40 (13238.650)
  CD19+CD5-, FU 85-PDFU 85, n=9 | -3911.67 (6060.974)
  CD19+CD5-, FU 169-PDFU 169, n=8 | -2170.38 (3568.904)

18. Secondary Outcome: Beta-2 Microglobulin at Cycle 1-Day 1
Description: Beta-2-microglobulin is a protein present on the surface of most cells. Higher levels indicate a poor prognosis of CLL. Beta-2 microglobulin was measured at Cycle 1-Day 1.
Time Frame: Cycle 1-Day 1
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Nanomoles per liter (NMOL/L)
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Nanomoles per liter (NMOL/L) | 301.442 (157.5521)

19. Secondary Outcome: Complement (CH50) at Cycle 1-Day 1 and Cycle 4-Day 85
Description: The CH50 is the serum complement to lyse 50% of sensitized red blood cells; it is a marker of complement activation. A high CH50 level suggests evidence for complement activation, whereas a low CH50 level suggests lack of complement activation. Peripheral blood samples were collected for analysis at Cycle 1-Day 1 and Cycle 4-Day 85.
Time Frame: Cycle 1-Day 1 and Cycle 4-Day 85
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects pPopulation.
Measure: Mean (Standard Deviation); unit: Kilo units per liter (KU/L)
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 10
Kilo units per liter (KU/L)
  Cycle 1-Day 1, n=10 | 42.63 (4.549)
  Cycle 4-Day 85, n=7 | 39.80 (5.791)

20. Secondary Outcome: Maximum (Peak) Plasma Concentration (Cmax) of Ofatumumab
Description: Maximum (peak) plasma drug concentration of ofatumumab was determined at Cycle 1-Day 1 and Cycle 3-Day 57. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr), and Cycle 3-Day 57 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr, 168 hr).
Time Frame: Cycle 1-Day 1 and Cycle 3-Day 57
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms/milliliter (µg/mL)
Groups:
- Overall Study Arm: ar. with previously untreated chronic lymphocytic leukemia (CLL) received intravenous (IV) infusions of ofatumumab on Day 1 (300 milligrams [mg]) and Day 8 (1000 mg) in the first cycle, followed by 1000 mg on the first day of each subsequent 28-day cycle in combination with oral chlorambucil 10 mg/meter squared (m^2) on Days 1-7 of each cycle for at least 3 cycles, until best overall response or up to 12 cycles. After the Treatment Phase (for par. in CR, PR or SD), survival and disease status were assessed 28 days after the first day of the last treatment cycle (Follow-up [FU] 1), 84 and 168 days after the day of FU1 (FU85 and FU169, respectively). For par. with disease progression (PD) during the Treatment Phase, post PD follow-up were done 28 days after the first day of the last treatment cycle (PDFU1) to assess safety. Survival status, date of next CLL therapy, and type of therapy were subsequently assessed 84 and 168 days after the day of PDFU1 (PDFU85 and PDFU169, respectively).
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 6
Micrograms/milliliter (µg/mL)
  Cycle 1-Day 1, n=6 | 59.4051 [43.125 to 81.831]
  Cycle 3-Day 57, n=5 | 296.1851 [197.449 to 444.295]

21. Secondary Outcome: Cmax of Serum Chlorambucil
Description: Cmax of serum chlorambucil was assesed at Cycle 1-Day 1, Cycle 1-Day 4 and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Ofatumumab +Chlorambucil: Par. with previously untreated chronic lymphocytic leukemia (CLL) received intravenous (IV) infusions of ofatumumab on Day 1 (300 milligrams [mg]) and Day 8 (1000 mg) in the first cycle, followed by 1000 mg on the first day of each subsequent 28-day cycle in combination with oral chlorambucil 10 mg/meter squared (m^2) on Days 1-7 of each cycle for at least 3 cycles, until best overall response or up to 12 cycles. After the Treatment Phase (for par. in CR, PR or SD), survival and disease status were assessed 28 days after the first day of the last treatment cycle (Follow-up [FU] 1), 84 and 168 days after the day of FU1 (FU85 and FU169, respectively). For par. with disease progression (PD) during the Treatment Phase, post PD follow-up were done 28 days after the first day of the last treatment cycle (PDFU1) to assess safety. Survival status, date of next CLL therapy, and type of therapy were subsequently assessed 84 and 168 days after the day of PDFU1 (PDFU85 and PDFU169, respectively).
Arm/Group | Ofatumumab +Chlorambucil
Number analyzed (Participants) | 6
ng/mL
  Cycle 1-Day 1, n=6 | 412.1241 [307.431 to 552.469]
  Cycle 1-Day 4, n=6 | 388.1516 [338.065 to 445.659]
  Cycle 3-Day 57, n=5 | 420.9367 [198.124 to 894.326]

22. Secondary Outcome: Cmax of Serum Phenyl Acetic Acid Mustard
Description: Cmax of chlorambucil metabolite phenyl acetic acid mustard was assesed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
ng/mL
  Cycle 1-Day 1, n=6 | 237.3587 [158.718 to 354.965]
  Cycle 1-Day 4, n=6 | 215.5603 [117.594 to 395.140]
  Cycle 3-Day 57, n=5 | 226.2480 [170.174 to 300.799]

23. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Ofatumumab
Description: Minimum plasma drug concentration of ofatumumab was determined at Cycle 1-Day 8, Cycle 2-Day 29, Cycle 3-Day 57, Cycle 4-Day 85, Cycle 5-Day 113, and Cycle 6-Day 141. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr), Cycle 2-Day 29 (pre-dose), Cycle 3-Day 57 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr, 168 hr), Cycle 4-Day 85 (pre-dose, 30 min post end of infusion), Cycle 5-Day 113 (pre-dose and end of infusion) and Cycle 6-Day 141 (pre-dose and end of infusion).
Time Frame: Cycle 1-Day 8, Cycle 2-Day 29, Cycle 3-Day 57, Cycle 4-Day 85, Cycle 5-Day 113, and Cycle 6-Day 141
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms/milliliter (µg/mL)
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Micrograms/milliliter (µg/mL)
  Cycle 1-Day 8, n=6 | 1.8693 [0.002 to 1779.832]
  Cycle 2-Day 29, n=4 | 73.0911 [59.023 to 90.511]
  Cycle 3-Day 57, n=5 | 57.8542 [15.444 to 216.724]
  Cycle 4-Day 85, n=4 | 82.1944 [24.517 to 275.563]
  Cycle 5-Day 113, n=4 | 98.3353 [44.749 to 216.089]
  Cycle 6-Day 141, n=4 | 82.9519 [25.286 to 272.123]

24. Secondary Outcome: Cmin of Chlorambucil
Description: Cmin of chlorambucil was assesed at Cycle 1-Day 4 and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 4 and Cycle 3-Day 57
Population: as for outcome 20
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
ng/mL
  Cycle 1-Day 4, n=6 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points.
  Cycle 3-Day 57, n=5 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points.

25. Secondary Outcome: Cmin of Phenyl Acetic Acid Mustard
Description: Cmin of chlorambucil metabolite phenyl acetic acid mustard was assesed at Cycle 1-Day 4 and Cycle 3-Day 57. Blood samples were collected at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 4 and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
ng/mL
  Cycle 1-Day 4, n=6 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points.
  Cycle 3-Day 57, n=5 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points.

26. Secondary Outcome: Total Plasma Clearance (CL) of Ofatumumab
Description: Plasma clearance is defined as the plasma volume which is totally cleared of drug per unit of time. Blood samples were collected at Cycle 1-Day1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr).
Time Frame: Cycle 1-Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Milliliters/hour (mL/hr)
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Milliliters/hour (mL/hr) | 172.64451 [46.4417 to 641.7962]

27. Secondary Outcome: Area Under the Drug Plasma Concentration-time Curve From Dosing to Time Tau (AUC[0-tau]) of Ofatumumab
Description: Area under the concentration time curve over the dosing interval (AUC[0-tau]) is a measure of drug exposure over time. AUC(0-tau) is defined as the area under the drug plasma/serum concentration-time curve from dosing to time tau, where tau is the length of the dosing interval of the drug. For ofatumumab it was assesed at Cycle 1-Day 1 and Cycle 3-Day 57. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr) and Cycle 3-Day 57 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr, 168 hr).
Time Frame: Cycle 1-Day 1 and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Hours*nanogram/milliliter (hr*ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Hours*nanogram/milliliter (hr*ng/mL
  Cycle 1-Day 1, n=6 | 1438.65082 [469.6310 to 4407.1120]
  Cycle 3-Day 57, n=5 | 62463.2072 [11630.9814 to 335453.399]

28. Secondary Outcome: AUC(0-tau) of Chlorambucil
Description: Area under the concentration time curve over the dosing interval (AUC[0-tau]) is a measure of drug exposure over time. AUC(0-tau) is defined as the area under the drug plasma/serum concentration-time curve from dosing to time tau, where tau is the length of the dosing interval of the drug. It was assesed at 1st (Cycle 1-Day 1), 4th (Cycle 1-Day 4), and 15th (Cycle 3-Day 57) chlorambucil administration. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Hr*ng/mL
  Cycle 1-Day 1, n=6 | 1191.17448 [871.1321 to 1628.7963]
  Cycle 1-Day 4, n=6 | 1060.28140 [714.1802 to 1574.1077]
  Cycle 3-Day 57, n=5 | 1259.26147 [662.4484 to 2393.7554]

29. Secondary Outcome: AUC(0-tau) of Phenyl Acetic Acid Mustard
Description: as for outcome 28
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Groups:
- Overall Study Arm: Par. with previously untreated chronic lymphocytic leukemia (CLL) received intravenous (IV) infusions of ofatumumab on Day 1 (300 milligrams [mg]) and Day 8 (1000 mg) in the first cycle, followed by 1000 mg on the first day of each subsequent 28-day cycle in combination with oral chlorambucil 10 mg/meter squared (m^2) on Days 1-7 of each cycle for at least 3 cycles, until best overall response or up to 12 cycles. After the Treatment Phase (for par. in CR, PR or SD), survival and disease status were assessed 28 days after the first day of the last treatment cycle (Follow-up [FU] 1), 84 and 168 days after the day of FU1 (FU85 and FU169, respectively). For par. with disease progression (PD) during the Treatment Phase, post PD follow-up were done 28 days after the first day of the last treatment cycle (PDFU1) to assess safety. Survival status, date of next CLL therapy, and type of therapy were subsequently assessed 84 and 168 days after the day of PDFU1 (PDFU85 and PDFU169, respectively).
Arm/Group | Overall Study Arm
Number analyzed (Participants) | 6
Hr*ng/mL
  Cycle 1-Day 1, n=6 | 1076.06435 [727.9702 to 1590.6069]
  Cycle 1-Day 4, n=6 | 984.02359 [608.0939 to 1592.3568]
  Cycle 3-Day 57, n=5 | 1038.87699 [799.7379 to 1349.5239]

30. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC[0-infinity]) for Ofatumumab
Description: The total AUC or AUC0-infinity is the area under the curve from time 0 extrapolated to infinite time. It was assesed on Cycle 1-Day 1. The samples were collected at Cycle 1-Day1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr).
Time Frame: Cycle 1-Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ug/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Hr*ug/mL | 1737.67475 [467.4381 to 6459.7075]

31. Secondary Outcome: AUC(0-infinity) for Chlorambucil
Description: The total AUC or AUC0-infinity is the area under the curve from time 0 extrapolated to infinite time. It was assesed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Hr*ng/mL
  Cycle 1-Day 1, n=6 | 1216.65216 [891.8548 to 1659.7349]
  Cycle 1-Day 4, n=6 | 1103.25854 [726.9103 to 1674.4561]
  Cycle 3-Day 57, n=5 | 1290.04709 [671.4967 to 2478.3764]

32. Secondary Outcome: AUC(0-infinity) for Phenyl Acetic Acid Mustard
Description: The total AUC or AUC(0-infinity) is the area under the curve from time 0 extrapolated to infinite time. It was assesed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Hr*ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
Hr*ng/mL
  Cycle 1-Day 1, n=6 | 1212.98123 [853.1396 to 1724.5987]
  Cycle 1-Day 4, n=6 | 1139.55544 [746.7799 to 1738.9147]
  Cycle 3-Day 57, n=5 | 1181.43279 [829.6354 to 1682.4058]

33. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Ofatumumab
Description: Volume of distribution at steady state (Vss) is defined as the distribution of a drug between plasma and the rest of the body at steady state. Samples were collected at Cycle 1-Day1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr).
Time Frame: Cycle 1-Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
mL | 5731.24330 [2746.3527 to 11960.2807]

34. Secondary Outcome: Plasma Half-life (t1/2) of Ofatumumab
Description: t1/2 is the time required for the plasma concentration of ofatumumab to decrease by half. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr) and Cycle 3-Day 57 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr, 168 hr).
Time Frame: Cycle 1-Day 1 and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 33.69818 [5.3514 to 212.1989]
  Cycle 3-Day 57, n=5 | 259.94722 [18.3504 to 3682.3409]

35. Secondary Outcome: Plasma Half-life (t1/2) of Chlorambucil
Description: t1/2 is the time required for the serum concentration of chlorambucil to decrease by half. Blood samples for serum concentration of chlorambucil was collected at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 1.06879 [0.8040 to 1.4209]
  Cycle 1-Day 4, n=6 | 1.74766 [1.2398 to 2.4636]
  Cycle 3-Day 57, n=5 | 1.38140 [1.0619 to 1.7971]

36. Secondary Outcome: Plasma Half-life (t1/2) of Phenyl Acetic Acid Mustard
Description: t1/2 is the time required for the plasma/serum concentration of phenylacetic acid mustard to decrease by half. Blood samples for serum concentration of phenylacetic acid mustard was collected at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 2.11378 [1.7689 to 2.5258]
  Cycle 1-Day 4, n=6 | 2.52918 [2.0358 to 3.1421]
  Cycle 3-Day 57, n=5 | 2.11552 [1.3110 to 3.4139]

37. Secondary Outcome: Time to Maximum Concentration (Tmax) of Ofatumumab
Description: Tmax is the time required for reaching maximum concentration of drug (Cmax). Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr) and Cycle 3-Day 57 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr, 168 hr).
Time Frame: Cycle 1-Day 1 and Cycle 3-Day 57
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 7.5400 [4.800 to 8.580]
  Cycle 3-Day 57, n=5 | 5.3200 [4.180 to 34.580]

38. Secondary Outcome: Time to Maximum Concentration (Tmax) of Chlorambucil
Description: Tmax is the time required for reaching maximum concentration of drug (Cmax). Blood samples were collected at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 2.9850 [1.530 to 6.000]
  Cycle 1-Day 4, n=6 | 1.9850 [0.470 to 4.150]
  Cycle 3-Day 57, n=5 | 3.0000 [1.450 to 3.980]

39. Secondary Outcome: Time to Maximum Concentration (Tmax) of Phenyl Acetic Acid Mustard
Description: as for outcome 38
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 3.9600 [2.030 to 6.000]
  Cycle 1-Day 4, n=6 | 3.4150 [1.420 to 5.950]
  Cycle 3-Day 57, n=5 | 3.9200 [1.970 to 5.930]

40. Secondary Outcome: Mean Residence Time to Infinity (MRTinf) of Ofatumumab
Description: MRTinf is the average amount of time that ofatumumab spends in the body. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr).
Time Frame: Cycle 1-Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours | 33.19679 [8.9888 to 122.6002]

41. Secondary Outcome: Mean Residence Time Inf (MRTinf) of Chlorambucil
Description: MRTinf is the average amount of time that chlorambucil spends in the body. Blood samples were collected at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 3.63147 [2.9689 to 4.4419]
  Cycle 1-Day 4, n=6 | 3.36698 [2.3904 to 4.7426]
  Cycle 3-Day 57, n=5 | 3.46924 [2.6156 to 4.6014]

42. Secondary Outcome: Mean Residence Time Inf (MRTinf) of Phenyl Acetic Acid Mustard
Description: MRTinf is the average amount of time that phenyl acetic acid mustard spends in the body. Blood samples were collected at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hours
  Cycle 1-Day 1, n=6 | 5.71852 [4.8439 to 6.7510]
  Cycle 1-Day 4, n=6 | 5.62096 [4.2681 to 7.4027]
  Cycle 3-Day 57, n=5 | 5.58632 [3.8972 to 8.0076]

43. Secondary Outcome: Volume of Distribution (Vz) of Ofatumumab
Description: Vz for ofatumumab was calculated as a ratio of the amount of ofatumumab in the body during the terminal phase to the plasma concentration during the terminal phase. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1hr, 2 hr, 24 hr, 72 hr, 120 hr).
Time Frame: Cycle 1-Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
mL | 8393.31979 [1691.3939 to 41650.7450]

44. Secondary Outcome: Apparent Total Clearance of the Drug From Plasma (CL/F) for Chlorambucil
Description: CL/F is defined as the apparent total clearance of the drug from plasma after oral administration of chlorambucil. It was assessed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr/m^2
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
L/hr/m^2
  Cycle 1-Day 1, n=6 | 8.21928 [6.0251 to 11.2126]
  Cycle 1-Day 4, n=6 | 9.06406 [5.9721 to 13.7569]
  Cycle 3-Day 57, n=5 | 7.75166 [4.0349 to 14.8921]

45. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Chlorambucil
Description: Vz/F of chlorambucil is defined as the apparent volume of distribution during terminal phase after non-intravenous (oral) administration of chlorambucil. It was assessed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: L/m^2
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
L/m^2
  Cycle 1-Day 1, n=6 | 12.67367 [8.2247 to 19.5291]
  Cycle 1-Day 4, n=6 | 22.85356 [14.9290 to 34.9846]
  Cycle 3-Day 57, n=5 | 15.44858 [9.2556 to 25.7853]

46. Secondary Outcome: %AUC_extrap of Ofatumumab
Description: %AUC_extrap is defined as the area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC. Samples were collected at Cycle 1-Day 1 (pre-dose, end of infusion, 10 min, 1 hr, 2 hr, 24 hr, 72 hr, 120 hr).
Time Frame: Cycle 1-Day 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUC after extrapolation
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
percentage of AUC after extrapolation | 3.99041 [0.4518 to 35.2433]

47. Secondary Outcome: %AUC_extrap of Chlorambucil
Description: %AUC_extrap is defined as the area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC. It was assessed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUC after extrapolation
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
percentage of AUC after extrapolation
  Cycle 1-Day 1, n=6 | 1.51853 [0.6086 to 3.7891]
  Cycle 1-Day 4, n=6 | 3.20042 [1.5963 to 6.4164]
  Cycle 3-Day 57, n=5 | 2.01046 [0.8604 to 4.6978]

48. Secondary Outcome: %AUC_extrap of Phenyl Acetic Acid Mustard
Description: as for outcome 47
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of AUC after extrapolation
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
percentage of AUC after extrapolation
  Cycle 1-Day 1, n=6 | 10.12009 [6.3465 to 16.1375]
  Cycle 1-Day 4, n=6 | 11.57955 [5.9445 to 22.5564]
  Cycle 3-Day 57, n=5 | 8.34549 [2.8229 to 24.6725]

49. Secondary Outcome: AUC (0-t) of Ofatumumab
Description: AUC (0-t) represents the area under the concentration curve of ofatumumab in plasma from 0 to time t hours. AUC (0-t) was assessed at 168 hours and 672 hours post-dose.
Time Frame: Cycle 1-Day 1 and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hr*µg/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hr*µg/mL
  AUC(0-168), Cycle 1-Day 1, n=6 | 1526.32835 [523.9756 to 4446.1580]
  AUC (0-672), Cycle 3-Day 57, n=5 | 58769.6326 [11273.1942 to 306378.977]

50. Secondary Outcome: AUC (0-t) of Chlorambucil
Description: AUC (0-t) represents the area under the concentration curve of chlorambucil in serum from 0 to time t hours. AUC (0-t) was assessed at 6 hours and 24 hours.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hr*ng/mL
  AUC(0-6), Cycle 1-Day 1, n=6 | 1069.26703 [811.5607 to 1408.8064]
  AUC(0-6), Cycle 1-Day 4, n=6 | 956.95261 [688.0559 to 1330.9359]
  AUC(0-6), Cycle 3-Day 57, n=5 | 1139.48401 [622.5013 to 2085.8169]
  AUC(0-24), Cycle 1-Day 1, n=6 | 1216.41085 [891.5347 to 1659.6721]
  AUC(0-24), Cycle 1-Day 4, n=6 | 1102.61367 [726.5937 to 1673.2279]
  AUC(0-24), Cycle 3-Day 57, n=5 | 1289.89389 [671.5260 to 2477.6795]

51. Secondary Outcome: AUC (0-t) of Phenyl Acetic Acid Mustard
Description: AUC (0-t) represents the area under the concentration curve of phenyl acetic acid mustard in serum from 0 to time t hours. AUC (0-t) was assessed at 6 hours and 24 hours.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hr*ng/mL
  AUC(0-6), Cycle 1-Day 1, n=6 | 755.55297 [459.9461 to 1241.1461]
  AUC(0-6), Cycle 1-Day 4, n=6 | 719.39401 [388.9287 to 1330.6493]
  AUC(0-6), Cycle 3-Day 57, n=5 | 743.47268 [568.9947 to 971.4531]
  AUC(0-24), Cycle 1-Day 1, n=6 | 1211.58911 [850.9549 to 1725.0600]
  AUC(0-24), Cycle 1-Day 4, n=6 | 1134.84945 [741.3620 to 1737.1855]
  AUC(0-24), Cycle 3-Day 57, n=5 | 1175.00443 [831.9658 to 1659.4858]

52. Secondary Outcome: Dose Normalized Cmax (Cmax/D) for Chlorambucil
Description: Cmax/D is defined as the maximum plasma concentration (Cmax) per unit dose. It was assessed at Cycle 1-Day 1, Cycle 1-Day 4 and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
ng/mL/mg
  Cycle 1-Day 1, n=6 | 26.49755 [17.9092 to 39.2044]
  Cycle 1-Day 4, n=6 | 24.95624 [21.0337 to 29.6103]
  Cycle 3-Day 57, n=5 | 28.82981 [15.0580 to 55.1973]

53. Secondary Outcome: Cmax/D for Phenyl Acetic Acid Mustard
Description: Cmax/D is defined as the maximum plasma concentration (Cmax) per unit dose. It was assessed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL/mg
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
ng/mL/mg
  Cycle 1-Day 1, n=6 | 15.26100 [9.5416 to 24.4087]
  Cycle 1-Day 4, n=6 | 13.85946 [7.0899 to 27.0926]
  Cycle 3-Day 57, n=5 | 15.49565 [12.5677 to 19.1057]

54. Secondary Outcome: AUC (0-6)/D, AUC(0-24)/D, AUC (0-inf)/D, and AUC (0-tau)/D of Chlorambucil
Description: Dose adjusted AUC for the indicated time points were assessed at Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57. In each sampling, blood samples were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr.
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL/mg
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hr*ng/mL/mg
  AUC(0-6)/D, Cycle 1-Day 1, n=6 | 68.74861 [50.6260 to 93.3586]
  AUC(0-6)/D, Cycle 1-Day 4, n=6 | 61.52734 [45.5317 to 83.1424]
  AUC(0-6)/D, Cycle 3-Day 57, n=5 | 78.04287 [43.5278 to 139.9265]
  AUC(0-24)/D, Cycle 1-Day 1, n=6 | 78.20923 [56.3038 to 108.6371]
  AUC(0-24)/D, Cycle 1-Day 4, n=6 | 70.89263 [48.0841 to 104.5204]
  AUC(0-24)/D, Cycle 3-Day 57, n=5 | 88.34439 [46.1690 to 169.0471]
  AUC(0-tau)/D, Cycle 1-Day 1, n=6 | 76.58665 [54.8550 to 106.9276]
  AUC(0-tau)/D, Cycle 1-Day 4, n=6 | 68.17087 [47.2363 to 98.3834]
  AUC(0-tau)/D, Cycle 3-Day 57, n=5 | 86.24639 [45.5445 to 163.3224]
  AUC(0-inf)/D, Cycle 1-Day 1, n=6 | 78.22474 [56.3280 to 108.6336]
  AUC(0-inf)/D, Cycle 1-Day 4, n=6 | 70.93409 [48.1052 to 104.5967]
  AUC(0-inf)/D, Cycle 3-Day 57, n=5 | 88.35489 [46.1675 to 169.0927]

55. Secondary Outcome: AUC (0-6)/D, AUC(0-24)/D, AUC (0-inf)/D and AUC (0-tau)/D of Phenyl Acetic Acid Mustard
Description: as for outcome 54
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: hr*ng/mL/mg
Arm/Group | Ofatumumab + Chlorambucil
Number analyzed (Participants) | 6
hr*ng/mL/mg
  AUC(0-6)/D, Cycle 1-Day 1, n=6 | 48.57834 [27.8596 to 84.7051]
  AUC(0-6)/D, Cycle 1-Day 4, n=6 | 46.25349 [23.9914 to 89.1730]
  AUC(0-6)/D, Cycle 3-Day 57, n=5 | 50.92019 [42.0701 to 61.6321]
  AUC(0-24)/D, Cycle 1-Day 1, n=6 | 77.89921 [49.8974 to 121.6154]
  AUC(0-24)/D, Cycle 1-Day 4, n=6 | 72.96523 [44.3328 to 120.0899]
  AUC(0-24)/D, Cycle 3-Day 57, n=5 | 80.47565 [53.4597 to 121.1442]
  AUC(0-tau)/D, Cycle 1-Day 1, n=6 | 69.18564 [43.0910 to 111.0825]
  AUC(0-tau)/D, Cycle 1-Day 4, n=6 | 63.26787 [36.8314 to 108.6797]
  AUC(0-tau)/D, Cycle 3-Day 57, n=5 | 71.15233 [53.3094 to 94.9674]
  AUC(0-inf)/D, Cycle 1-Day 1, n=6 | 77.98872 [50.0093 to 121.6221]
  AUC(0-inf)/D, Cycle 1-Day 4, n=6 | 73.26780 [44.6278 to 120.2876]
  AUC(0-inf)/D, Cycle 3-Day 57, n=5 | 80.91593 [53.1321 to 123.2284]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment until follow-up for survival (up to Week 62.3).
Description: SAEs and non-serious AEs are reported for members of the All Subjects Population, comprised of all participants who received at least one dose of investigational product.
Groups:
- Ofatumumab+Chlorambucil: Participants with previously untreated chronic lymphocytic leukemia (CLL) received intravenous (IV) infusions of ofatumumab on Day 1 (300 milligrams [mg]) and Day 8 (1000 mg) in the first cycle, followed by 1000 mg on the first day of each subsequent 28 day cycle in combination with chlorambucil 10 mg/meter squared (m^2) orally on Days 1-7 of every 28 day cycle for a minimum of 3 cycles, until best overall response or a maximum of 12 cycles. After completion of the Treatment Phase (for participants in CR, PR or SD), survival and disease status assessment visits were performed 28 days after the first day of the last treatment cycle (Follow-up [FU] 1), 84 days, and 168 days after the day of FU 1 (FU 85 and FU 169, respectively). For participants experiencing disease progression during the Treatment Phase, the post progressive disease (PD) follow-up for safety assessments were performed 28 days after the first day of the last treatment cycle (PDFU 1). Subsequent follow-up was performed 8
Arm/Group | Ofatumumab+Chlorambucil
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab+Chlorambucil (N=10)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab+Chlorambucil (N=10)
White blood cell count decreased (Investigations) | 5
Neutrophil count decreased (Investigations) | 4
Platelet count decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 2
Amylase increased (Investigations) | 1
Beta 2 microglobulin increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Blood potassium increased (Investigations) | 1
Blood sodium decreased (Investigations) | 1
Electrocardiogram ST segment depression (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 3
Chills (General disorders) | 2
Oedema (General disorders) | 2
Chest discomfort (General disorders) | 1
Malaise (General disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Nasopharyngitis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Insomnia (Psychiatric disorders) | 2
Palpitations (Cardiac disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.